CLINICAL TRIAL: NCT06352099
Title: Evaluation of Dietary Supplementation With Hesperidin and Proanthocyanidins on Cognitive and Motor Functions in Elderly Subjects
Brief Title: Dietary Supplementation and Cognitive Functions in the Elderly
Acronym: ESPINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 6315
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Impairment; Old Age; Debility
Keywords: Elderly; Cognitive performance; Fatigue; Quality of life; Falls; Nutraceutical
MeSH Terms: conditions — Cognitive Dysfunction; Frailty; Fatigue | interventions — Dietary Supplements; Hesperidin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G-Alt12 (Experimental): G-Alt12 patients, without making any changes to their current drug routine, will take 1 stick per day of Altemor® for 8 weeks, go for a period of 4 weeks without taking the food supplement, and then take 2 sticks per day of Altemor® for another 8 weeks.
  Interventions: Dietary Supplement: Dietary supplement with micronised diosmin, hesperidin and herbal extracts
- G-Alt21 (Experimental): G-Alt21 patients, without making any changes to their current medication routine, will take 2 sticks per day of Altemor® for 8 weeks, do a 4-week period without taking the dietary supplement, and then take 1 stick per day of Altemor® for another 8 weeks.
  Interventions: Dietary Supplement: Dietary supplement with micronised diosmin, hesperidin and herbal extracts
- G-Con (No Intervention): G-Con patients will undergo clinical and instrumental evaluations at the study endpoints

INTERVENTIONS:
Dietary Supplement: Dietary supplement with micronised diosmin, hesperidin and herbal extracts — Taking a dietary supplement with micronised diosmin, hesperidin and plant extracts 1 or 2 sticks per day, as per the study design.
  Other Names: Altemor®
  Arms: G-Alt12; G-Alt21

SUMMARY:
In recent years, globally, there has been a growth in both the size and the proportion of older adults in the world population. The World Health Organization (WHO) has estimated that by 2030, 1 in 6 people will be 60 years of age or older, and that by 2050, the population of older adults will reach 2.1 billion. The population of older adults (over 80 years) will triple to 426 million by 2050. In particular, Italy represents the second country with the oldest population in the world.

Age-related evolution is a gradual and continuous process involving a series of physical and cognitive changes, which, however, has no real 'onset' age. In fact, rather than chronological age, the concept of 'elderly' is based on the individual's degree of self-sufficiency and independence. From a biological point of view, ageing is the set of changes at the molecular and cellular level that occur over time and lead to multi-system functional impairment. It is a process directly related to frailty, falls, and disability.

An important factor in counteracting frailty is nutritional intake. Humans ingest approximately 500 g of chemical compounds daily through their diet, most of which are components of plants or vegetables in general. In addition to the well-known macronutrients (proteins, fats, and carbohydrates) and micronutrients (minerals and vitamins), the plant world provides other elements, such as phenols, terpenes, terpenoids, alkaloids, purines, pyrimidines, nucleic acids, and steroids, that exert powerful biological activities. These components are generically called phytochemicals. Epidemiological studies have established that diets rich in plant-based foods help prevent many diseases, such as cardiovascular, metabolic, neurovegetative, and inflammatory diseases.

Phytochemical compounds are an extremely diverse set of elements that, when taken at significant levels, have a protective effect on human health. These substances exert various biological functions, such as antioxidant activity, modulation of detoxifying enzymes, stimulation of the immune system, reduction of platelet aggregation, modulation of hormone metabolism, reduction of blood pressure, and antibacterial and antiviral activity.

Among the phytochemical compounds, flavonoids represent a category of polyfunctional substances with high bioactivity, comprising more than 5000 compounds. They possess biochemical properties of functional interest in the nutritional and therapeutic fields; for example, rutin, diosmin, and hesperidin are present in some pharmaceutical specialties; flavonoids from ginkgo biloba, hawthorn, and red vine are the main components of many phytotherapeutic extracts. Flavonoids have been shown to play an important role in cardioprotection. Furthermore, in neuroprotection, anthocyanin-rich fruits play a protective role against age-related decline in cognitive functions.

However, few studies have evaluated the effect of hesperidin and proanthocyanidins on motor, cognitive, and functional aspects in the elderly.

Altemor® is a food supplement based on micronized diosmin, hesperidin, and herbal extracts that has an important integrative supporting action in optimising blood microcirculation.

The aim of the study is to evaluate the contribution of dietary supplementation with Altemor® on cognitive function, balance, fatigue, and some domains of quality of life in elderly subjects.

DETAILED DESCRIPTION:
Thirty-six patients evaluated and treated at the UOS Post-Acute Rehabilitation, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, who meet the inclusion criteria, will be recruited. Patients will be divided into three groups by randomization, as specified below. One group (G-Alt12), without any modification of the current pharmacological routine, will take 1 stick per day of Altemor® for 8 weeks, do 4 weeks of wash-out, and then take 2 sticks per day of Altemor® for another 8 weeks; the other group (G-Alt21), without any modification of the current pharmacological routine, will take 2 sticks per day of Altemor® for 8 weeks, do 4 weeks of wash-out, and then take 1 stick per day of Altemor® for another 8 weeks. The third group (G-con), without any modification of the current drug routine, if any, will not take Altemor® but will only be evaluated according to the endpoints in the study and described below.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 32 kg/m2
* Non-smoker
* Cognitive ability to carry out simple orders and to understand the physiotherapist's instructions [assessed by the Mini Mental State Examination (correct score between 22 and 27)]
* Independence in instrumental activities of daily living [assessed by the Instrumental Activities of Daily Living (score < 5)
* Medication stability of at least 12 months for taking any medication for hypertension, hyperlipidemia, inflammation, hypercholesterolemiaand hypercoagulation;
* Ability to walk independently or with little assistance;
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Previous history of stroke and/or myocardial infarction;
* Presence of altered mood [assessed by the Hospital Anxiety and Depression Scale (score ≤ 8)].
* Presence of kidney or intestinal disease, pancreatitis, diabetes or any other endocrine disorder
* Presence of demyelinating and dysmyelinating diseases;
* Presence of anticoagulant or antiplatelet drugs;
* Systemic, neurological or cardiac diseases that make walking unsafe or cause motor deficits;
* Oncological pathologies;
* Vegetarian diet, regular intake of supplements including fish oil, fatty acids, vitamins and minerals
* Orthopaedic or postural problems;
* Presence of plantar ulcers;
* Partial or total amputation of foot segments.
* Inability to provide informed consent.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Trial Making Test (TMT) | Change from Baseline TMT at 8 and 16 weeks
  The TMT measures flexibility of thinking on a visual-motor sequencing task. It consists of two parts, A and B, where 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.).
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
  Trail A: Average 29 seconds, Deficient > 78 seconds, Rule of Thumb Most in 90 seconds Trail B: Average 75 seconds, Deficient > 273 seconds, Rule of Thumb Most in 3 minutes

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change from Baseline SPPB at 8 and 16 weeks
  SPPB is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). Three domains, which include balance, usual or self-selected gait speed, and lower limb strength, are assessed by a three-stage balance test (feet side-by-side, semitandem, and tandem positions), a 3-m or 4-m gait speed test (time spent to walk the course), and a repetitive chair stand test (five times chair sit-to-stand test), respectively. A 0- to 12-point scale is used to score the sum of the three assessments with higher point values corresponding with greater levels of physical function and lower disability, whereas lower point values correspond with lower levels of physical function and higher disability, respectively.
HandGrip Strenght Test (HGST) | Change from Baseline HGST at 8 and 16 weeks
  HGST is a test performed with a dynamometer, which goes to assess muscle strength (in kilograms). Starting with the elbow flexed to 90°, the patient must squeeze the dynamometer as hard as they can at one time. Three repeated measurements are taken on each side 20 seconds apart.
  The average of the three assessments is used as the final value.
Silver Index (SI) | Change from Baseline SI at 8 and 16 weeks
  The SI is an objective test to identify the risk of falling, which is carried out using the Hunova robotic platform. It consists of seven domains:
  (i) static balance (ii) dynamic balance (iii) reactive balance (iv) sensory integration (v) stability limits (vi) sitting-to-standing position (vii) gait speed.
  At the end of the evaluation you get a percentage that indicates the risk of falling
Mental Deterioration battery (MDB) | Change from Baseline MDB at 8 and 16 weeks
  The MDB is a neuropsychological test battery for detecting mental deterioration and comprises 7 tests divided into verbal and visuospatial tests, which can be administered independently of each other.
  VERBAL TESTS are: immediate and delayed recall of Rey's 15 words, phonological verbal fluency; sentence construction VISUAL-SPACE TESTS are: Raven's coloured progressive matrices (PM47; immediate visual memory; copying of freehand drawings)
  All MDB tests are corrected using the Equivalent Scores method, after correction for factors (age, years of schooling) of the score obtained.
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline HADS at 8 and 16 weeks
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale, the score is the sum of the respective seven items (ranging from 0 to 21).
  The two sub-scales, anxiety and depression, have been found to be independent measures. In its current form, the HADS is now divided into four stages:
  Scores of:
  0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)
EuroQol- 5 Dimension (EQ-5D) | Change from Baseline EQ-5D at 8 and 16 weeks
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.
Modified Fatigue Impact Scale (MFIS) | Change from Baseline MFIS at 8 and 16 weeks
  The MFIS is an instrument that provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items while the abbreviated version has 5 items.
  The MFIS is a structured, self-report questionnaire that the patient can generally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument.
  The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Giovannini, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giovannini S, Lauria A, Malizia AM, Lama E, Morciano N, Biscotti L, Loreti C, Castelli L. The Effectiveness of Hesperidin, Diosmin and Proanthocyanidins Nutritional Supplementation on Cognitive and Motor Functions in Older Adults: A Pilot Randomized Control Study. J Am Nutr Assoc. 2026 Jan;45(1):24-36. doi: 10.1080/27697061.2025.2526600. Epub 2025 Jul 22. PMID 40694049